CLINICAL TRIAL: NCT00685841
Title: A Double-Blind, Double-Dummy, Randomized, Placebo- and Active-Controlled, Multicenter, Parallel-Group Study of (R,R)-Formoterol in the Treatment of Subjects With Chronic Obstructive Pulmonary Disease
Brief Title: A Pivotal Study of the Safety and Effectiveness of Arformoterol in Subjects With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 091-050
Record Dates: First submitted 2008-05-23; First posted 2008-05-28 (Estimated); Last update posted 2012-11-02 (Estimated); Status verified 2012-11

CONDITIONS: COPD
Keywords: Chronic obstructive pulmonary disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Formoterol Fumarate; Salmeterol Xinafoate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- A (Experimental): Arformoterol 50 mcg QD and placebo MDI
  Interventions: Drug: Arformoterol tartrate inhalation solution
- B (Experimental): Arformoterol 25 mcg BID and placebo MDI
  Interventions: Drug: Arformoterol tartrate inhalation solution
- C (Experimental): Arformoterol 15 mcg BID and placebo MDI
  Interventions: Drug: Arformoterol tartrate inhalation solution
- D (Active Comparator): Salmeterol MDI 42 mcg BID and placebo inhalation solution
  Interventions: Drug: Salmeterol MDI
- E (Placebo Comparator): Placebo BID MDI and inhalation solution
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Arformoterol tartrate inhalation solution — Arformoterol 50 mcg QD
  Other Names: (R,R-)formoterol; Brovana
  Arms: A
Drug: Arformoterol tartrate inhalation solution — Arformoterol 25 mcg BID
  Other Names: (R,R)-formoterol; Brovana
  Arms: B
Drug: Arformoterol tartrate inhalation solution — Arformoterol 15 mcg BID
  Other Names: (R,R)-formoterol; Brovana
  Arms: C
Drug: Salmeterol MDI — Salmeterol MDI 42 mcg BID
  Other Names: Serevent
  Arms: D
Drug: Placebo — Placebo BID MDI
  Arms: E

SUMMARY:
A 12 week study to investigate the safety and effectiveness of arformoterol given twice daily compared to placebo in subjects with COPD.

DETAILED DESCRIPTION:
This study is a double-blind, double-dummy, randomized, placebo- and active-controlled, multicenter, parallel-group study of adult subjects with a primary clinical diagnosis of COPD. Approximately 800 subjects were to be randomized in this study. Study participation consisted of a total of eight (8) study visits over approximately four (4) months for each subject. This study was previously posted by Sepracor Inc. In October 2009, Sepracor Inc. was acquired by Dainippon Sumitomo Pharma., and in October 2010, Sepracor Inc's name was changed to Sunovion Pharmaceuticals Inc.

ELIGIBILITY:
Inclusion Criteria

* Subject may be male or female and must be aged less than or equal to 35 years on the day the informed consent is signed.
* Female subjects greater than or equal to 65 years of age must have a serum pregnancy test conducted at Visit 1 and confirmed negative prior to randomization. Subjects of childbearing potential must be using an acceptable method of birth control.
* Female subjects who are considered not of childbearing potential must be:

  * documented surgically sterile (defined as status post-hysterectomy or bilateral tubal ligation) OR
  * postmenopausal
* Subject must have a primary diagnosis of COPD, which may include components of chronic bronchitis and/or emphysema. Diagnosis can be made during the screening process.
* Subject must have a minimum smoking history of 15 pack-years (pack-years = the number of cigarette packs per day times the number of years).
* Subject must have a chest x-ray that is consistent with the diagnosis of COPD (e.g., not diagnostic of pneumonia, other infection, atelectasis, or pneumothorax or other active/ongoing pulmonary conditions) and taken less than or equal to 3 months prior to study start. If there is no chest x-ray taken less than or equal to 3 months prior to study start, or if recent results are unavailable for review, a chest x-ray will be performed.
* Subject must be able to complete all study questionnaires and logs reliably. Exclusion Criteria
* Female subject who is pregnant or lactating.
* Subject who has participated in an investigational drug study within 30 days prior to study start, or who is currently participating in another investigational drug study.
* Subject whose schedule or travel prevents the completion of all required visits.
* Subject who is scheduled for in-patient hospitalization, including elective surgery (in patient or out-patient) during the trial.
* Subject with life-threatening/unstable respiratory status, including upper or lower respiratory tract infection, within the previous 30 days prior to study start.
* Subject with a known history of asthma or any chronic respiratory disease (including a current history of sleep apnea) other than COPD (chronic bronchitis and/or emphysema).
* Subject with a history of cancer except non-melanomatous skin cancer. Subjects with a history of cancer that is considered surgically cured and without a recurrence within the past 10 years may participate in the study. History of hematologic/lymphatic malignancy treated with chemotherapy or radiation is not allowed.
* Subject with a history of lung resection of more than one full lobe.
* Subject who requires continuous supplemental oxygen therapy (unless subject resides at elevation greater than or equal to 4,000 feet).
* Subject who has had a change in dose or type of any medications for COPD within 14 days prior to the screening visit.
* Subject with a known sensitivity to (R,R)-formoterol, ipratropium, salmeterol or albuterol or any of the excipients contained in any of these formulations.
* Subject with a history of substance abuse or drug abuse within 12 months of study start, or with a positive urine drug screen at study start.
* Subject using any prescription drug for which concomitant beta-agonist administration is contraindicated (e.g., beta-blockers).

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 717 (Actual)
Dates: Start 2002-02; Primary Completion 2003-06 (Actual); Study Completion 2003-06 (Actual)

PRIMARY OUTCOMES:
Percent change from study baseline FEV1 to the end of the dosing interval (12 hours post-second dose for the BID treatment arms and 24 hours post-dose for the QD treatment arm) | Weeks -2, 0, 3, 6, 9, 12

SECONDARY OUTCOMES:
Time-normalized area under the percent change from visit pre-dose curve for FEV1 over 12 hours (nAUC0-12) | Weeks -2, 0, 3, 6, 9, 12
Peak percent of predicted FEV1 | Weeks -2, 0, 3, 6, 9, 12
Time-normalized area under the percent change from study baseline curve for FEV1 over 12 hours (nAUC0-12) | Weeks -2, 0, 3, 6, 9, 12
Time-normalized area under the percent change from study baseline curve for FEV1 over 24 hours (nAUC0-24) | Weeks -2, 0, 3, 6, 9, 12
Timepoint changes in FEV1 | Weeks -2, 0, 3, 6, 9, 12
Time to onset of response | Weeks -2, 0, 3, 6, 9, 12
Time to peak change in FEV1 | Weeks -2, 0, 3, 6, 9, 12
At-home and in-clinic peak expiratory flow rate (PEFR) | Weeks -2, 0, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12
Ipratropium bromide MDI use | Weeks -2, 0, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12
Racemic albuterol MDI use | Weeks -2, 0, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12
Exacerbations of COPD | Weeks -2, 0, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12
COPD symptom ratings (over 12 weeks of treatment) | Weeks -2, 0, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12
Relationship between plasma concentrations of (R,R) formoterol and selected pharmacodynamic parameters | Weeks -2, 0, 3, 6, 9, 12

CONTACTS AND LOCATIONS:
Locations (52):
- United States (52):
  - Anniston, Alabama
  - Birmingham, Alabama
  - Jasper, Alabama
  - Mobile, Alabama
  - Oxford, Alabama
  - Little Rock, Arkansas
  - Los Angeles, California
  - Mirage, California
  - Mission Hills, California
  - San Diego, California
  - Santa Ana, California
  - Signal Hill, California
  - Colorado Springs, Colorado
  - Denver, Colorado
  - Wheat Ridge, Colorado
  - Clearwater, Florida
  - DeLand, Florida
  - Miami, Florida
  - Ocala, Florida
  - Pensacola, Florida
  - St. Petersburg, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Austell, Georgia
  - Decatur, Georgia
  - Bloomington, Illinois
  - Evansville, Indiana
  - Shawnee Mission, Kansas
  - Minneapolis, Minnesota
  - Charles, Missouri
  - Las Vegas, Nevada
  - Margate City, New Jersey
  - South Bound Brook, New Jersey
  - Albuquerque, New Mexico
  - Endwell, New York
  - Ithaca, New York
  - New York, New York
  - Charlotte, North Carolina
  - Raleigh, North Carolina
  - Spartanburg, North Carolina
  - Wilmington, North Carolina
  - Cincinnati, Ohio
  - Tulsa, Oklahoma
  - Medford, Oregon
  - Pittsburgh, Pennsylvania
  - Charleston, South Carolina
  - Houston, Texas
  - Irving, Texas
  - San Antonio, Texas
  - Chesapeake, Virginia
  - Richmond, Virginia
  - Tacoma, Washington